CLINICAL TRIAL: NCT03859557
Title: The Evaluation of Patients With Esophageal and Foregut Disorders With WATS (Wide Area Transepithelial Sample With 3-Dimensional Computer-Assisted Analysis) vs. 4-Quadrant Forceps Biopsy
Status: Completed | Type: Observational
Sponsor: CDx Diagnostics (Industry)
Collaborators: Foundation for Surgical Innovation and Education (Unknown)
Responsible Party: Principal Investigator, Steven DeMeester, MD, President and Executive Director The Foundation for Research and Education in Esophageal and Foregut Disease, The Oregon Clinic
Other Study IDs: CDx 810b
Record Dates: First submitted 2019-02-15; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: GERD; Barrett Esophagus; Low Grade Esophageal Glandular Dysplasia; Esophageal Diseases
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus; Esophageal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 4-Quadrant Random Forceps Biopsy: Random sampling within a quadrant of esophageal tissue using forceps.
- WATS biopsies: Wide area transepithelial sampling with computer aided pathologic interpretation of tissue.

SUMMARY:
Patients scheduled to undergo routine upper endoscopy for foregut or esophageal symptoms or undergoing surveillance for Barrett's esophagus with no dysplasia or low-grade dysplasia are candidates for participation, but patients with known high-grade dysplasia or adenocarcinoma or with a history of prior endoscopic resection or ablation for these conditions are not candidates for participation.

At endoscopy, all patients will be initially assessed for the presence of an endoscopic suspicious lesion using white light and if appropriate narrow band imaging or similar enhanced imaging techniques. All suspicious lesions undergo targeted biopsy first, and then either 4-Quadrant Random Forceps Biopsy or WATS biopsies of the GEJ and if present the columnar-lined esophagus based on the assigned randomization away from the area of targeted biopsies. A biopsy will be obtained from the antrum in each patient to assess for H. pylori infection and the presence of intestinal metaplasia.

DETAILED DESCRIPTION:
Patients scheduled to undergo routine upper endoscopy for foregut or esophageal symptoms will be enrolled. Patients undergoing surveillance for Barrett's esophagus with no dysplasia or low-grade dysplasia are candidates for participation, but patients with known high-grade dysplasia or adenocarcinoma or with a history of prior endoscopic resection or ablation for these conditions are not candidates for participation. Informed consent will be obtained from every patient prior to enrollment.

Patients will be randomized prior to starting the procedure. Each patient will receive a randomization code at the time of randomization. It is important that the randomization code be included in the Case Report Form submitted with each patient, and will represent the unique deidentified code for each patient's data for inclusion in the study database.

At endoscopy, all patients will be initially assessed for the presence of an endoscopic suspicious lesion using white light and if appropriate narrow band imaging or similar enhanced imaging techniques. All suspicious lesions undergo targeted biopsy first, and then either 4-Quadrant Random Forceps Biopsy or WATS biopsies of the GEJ and if present the columnar-lined esophagus based on the assigned randomization away from the area of targeted biopsies. A biopsy will be obtained from the antrum in each patient to assess for H. pylori infection and the presence of intestinal metaplasia.

Targeted forceps biopsies of any endoscopic suspicious area will be placed in a separate pathology bottle from those obtained from 4-Quadrant Random Forceps Biopsy and analyzed separately as well.

All the components needed to perform WATS biopsies are included in a kit with complete written instructions.

WATS specimens will be analyzed by CDx Diagnostics. Investigator will ship the WATS specimens to CDx Diagnostics in accordance with CDx's instructions. Forceps biopsies will be analyzed by institution's pathology department and the pathology department of each additional site participating in the Study per standard protocol.

The Investigator will determine appropriate follow-up of patients with and without IM or dysplasia detected by WATS or FB per standard individual and / or institution protocol.

Investigator and all investigators at the additional sites will supply the study coordinator with de-identified data for each specimen, such de-identified data including patient demographics, endoscopic findings, and results of the FB of GEJ, antrum plus / minus esophagus. Study Data will be maintained on a secure database by the study coordinator during the Term and for six years thereafter.

Biopsies with intestinal metaplasia or dysplasia may be reviewed by a central pathologist to confirm the original pathologic interpretation when there is a discrepancy between WATS and FB that is greater than 10%.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females at least 18 years of age undergoing routine upper endoscopy to evaluate symptoms of esophageal or foregut disorders (reflux disease, BE, esophageal strictures, swallowing disorders, dyspepsia, hiatal hernias, motility issues, gastric issues).
* Institutional Review Board (IRB)-approved consent must be signed by patients prior to participating in this study.

Exclusion Criteria:

* Patients who do not undergo either FB or WATS biopsy
* Patients with inadequate WATS or FB specimens
* Known history of high-grade dysplasia or adenocarcinoma
* Prior history of endoscopic resection or ablation for Barrett's with high-grade dysplasia or adenocarcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are those who undergo routine upper endoscopy while under sedation to evaluate foregut or esophageal symptoms.
Sampling Method: Probability Sample
Enrollment: 1032 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Yield of WATS biopsies compared to Forceps biopsies | 12 months
  Intestinal metaplasia is a premalignant change in the normal epithelium lining the esophagus and gastroesophageal junction. It is evaluated on tissue samples from these areas by a pathologist under a microscope, who then determines if intestinal metaplasia is present or not. All specimens retrieved by upper endoscopy, whether by standard biopsy or by WATS, will be examined by a pathologist. The pathology reports will be reviewed and the frequency that intestinal metaplasia is found by standard biopsy vs WATS will be statistically compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

REFERENCES:
- [Derived] DeMeester S, Smith C, Severson P, Loveitt A, Jobe B, Woodworth P, Wilcox D, Dunst C; Hawaii Esophageal Course Study Group. Multicenter randomized controlled trial comparing forceps biopsy sampling with wide-area transepithelial sampling brush for detecting intestinal metaplasia and dysplasia during routine upper endoscopy. Gastrointest Endosc. 2022 Jun;95(6):1101-1110.e2. doi: 10.1016/j.gie.2021.11.044. Epub 2021 Dec 10. PMID 34902373